CLINICAL TRIAL: NCT03974100
Title: A Randomized, Double-blind, Multicenter Integrated Phase I/III Study in Postmenopausal Women With Osteoporosis to Compare the Pharmacokinetics, Pharmacodynamics, Efficacy, Safety and Immunogenicity of GP2411 (Proposed Biosimilar Denosumab) and Prolia® (EU-authorized)
Brief Title: Study Investigating PK, PD, Efficacy, Safety, and Immunogenicity of Biosimilar Denosumab (GP2411) in Patients With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGP24112301; 2018-003523-11 (EudraCT Number); NCT03991338 (obsolete NCT alias)
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Postmenopausal Women With Osteoporosis
Keywords: Prolia; GP2411; denosumab; postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GP2411 (Experimental): 60 mg /mL subcutaneous injection every 6 months
  Interventions: Biological: GP2411
- EU authorized Prolia (Active Comparator): 60 mg /mL subcutaneous injection every 6 months
  Interventions: Biological: EU-Prolia (EU-authorized Prolia®)

INTERVENTIONS:
Biological: GP2411 — 60 mg /mL subcutaneous injection every 6 months
  Arms: GP2411
Biological: EU-Prolia (EU-authorized Prolia®) — 60 mg /mL subcutaneous injection every 6 months
  Arms: EU authorized Prolia

SUMMARY:
This study was conducted to assess if there were any clinically meaningful differences in pharmacokinetics (PK), pharmacodynamics (PD), efficacy, safety, or immunogenicity between GP2411 (proposed biosimilar denosumab) and EU-authorized Prolia® (denosumab).

DETAILED DESCRIPTION:
This was an international, multicenter, randomized, double-blind, parallel-group study with a total duration of up to 83 weeks.

The study comprised a screening period of up to 5 weeks to assess a subject's eligibility and two treatment periods: Treatment Period 1 (TP1) from Day 1 to Week 52 and Treatment Period 2 (TP2) from Week 52 to Week 78.

Women with postmenopausal osteoporosis (PMO) were randomized on Day 1 in a 1:1 ratio to receive either two 60 mg subcutaneous (s.c.) doses at 26-week intervals of GP2411 (proposed biosimilar denosumab) or EU-Prolia (EU-authorized Prolia®) during TP1. At Week 52, participants in the EU-Prolia group were re-randomized 1:1 to either continue with a third dose of EU-Prolia or switch to GP2411 for TP2. Participants in the GP2411 group continued the treatment with a third dose of GP2411 in TP2. The End of Study was achieved at Week 78.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, diagnosed with osteoporosis
* Aged ≥ 55 and ≤ 80 years at screening
* Body weight ≥ 50 kg and ≤ 90 kg at screening
* Absolute bone mineral density consistent with T-score ≤ -2.5 and ≥ -4.0 at the lumbar spine as measured by DXA
* At least two vertebrae in the L1-L4 region and at least one hip joint are evaluable by DXA

Exclusion Criteria:

* Previous exposure to denosumab (Prolia, Xgeva, or biosimilar denosumab)
* History and/or presence of one severe or more than two moderate vertebral fractures or hip fracture
* History and/or presence of bone metastases, bone disease or metabolic disease
* Ongoing use of any osteoporosis treatment or use of prohibited treatment
* Other bone active drugs
* History and/or current hypoparathyroidism or hyperparathyroidism, hypocalcemia or hypercalcemia

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women, diagnosed with osteoporosis
Enrollment: 527 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (6):
  - Sandoz Investigational Site, Peoria, Arizona
  - Sandoz Investigational Site, Miami, Florida
  - Sandoz Investigational Site, Wichita, Kansas
  - Sandoz Investigational Site, Duncansville, Pennsylvania
  - Sandoz Investigational Site, Wyomissing, Pennsylvania
  - Sandoz Investigational Site, Carrollton, Texas
- Bulgaria (2):
  - Sandoz Investigational Site, Plovdiv
  - Sandoz Investigational Site, Sofia
- Czechia (8):
  - Sandoz Investigational Site, Ostrava, Czech Republic
  - Sandoz Investigational Site, Hradec Králové, CZE
  - Sandoz Investigational Site, Brno
  - Sandoz Investigational Site, Ostrava
  - Sandoz Investigational Site, Pardubice
  - Sandoz Investigational Site, Pilsen
  - Sandoz Investigational Site, Prague
  - Sandoz Investigational Site, Uherské Hradiště
- Japan (5):
  - Sandoz Investigational Site, Fujimi, Saitama
  - Sandoz Investigational Site, Chuoh-ku, Tokyo
  - Sandoz Investigational Site, Hachiōji, Tokyo
  - Sandoz Investigational Site, Kiyose, Tokyo
  - Sandoz Investigational Site, Shinagawa, Tokyo
- Poland (7):
  - Sandoz Investigational Site, Krakow, Lesser Poland Voivodeship
  - Sandoz Investigational Site, Bialystok
  - Sandoz Investigational Site, Bydgoszcz
  - Sandoz Investigational Site, Lodz
  - Sandoz Investigational Site, Nadarzyn
  - Sandoz Investigational Site, Torun
  - Sandoz Investigational Site, Warsaw
- Spain (6):
  - Sandoz Investigational Site, Santiago de Compostela, A Coruna
  - Sandoz Investigational Site, Sabadell, Barcelona
  - Sandoz Investigational Site, Santiago de Compostela, Galicia
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Madrid
  - Sandoz Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 43 investigative sites in 6 countries.
Pre-assignment Details: The screening period of up to 5 weeks began after the subject had provided written informed consent and ended at the randomization visit (Day 1). On Day 1, participants were randomized in a 1:1 ratio to receive either GP2411 or EU-Prolia during Treatment Period 1 (TP1).
  At Week 52, participants in the EU-Prolia group were re-randomized 1:1 to either continue with EU-Prolia or switch to GP2411 for Treatment Period 2 (TP2). Participants in the GP2411 group continued with GP2411 for TP2.
Groups:
- GP2411: Two 60 mg s.c. doses at 26-week intervals of GP2411 (proposed biosimilar denosumab) in TP1
- EU-Prolia: Two 60 mg s.c. doses at 26-week intervals of EU-Prolia (denosumab) in TP1
- GP2411/GP2411: Participants treated with GP2411 in TP1 continued with a third dose of GP2411 in TP2
- EU-Prolia/EU-Prolia: Participants treated with EU-Prolia in TP1 were re-randomized to continue with a third dose of EU-Prolia in TP2
- EU-Prolia/GP2411: Participants treated with EU-Prolia in TP1 were re-randomized to switch to GP2411 in TP2
Period: TP1 - Day 1 to Week 52
Arm/Group | GP2411 | EU-Prolia | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Started | 263 | 264 | 0 | 0 | 0
Per-Protocol Set (PPS) | 233 | 230 | 0 | 0 | 0
TP1 Full Analysis Set (TP1 FAS) | 255 | 257 | 0 | 0 | 0
Pharmacodynamic Analysis Set (PDS) | 228 | 213 | 0 | 0 | 0
Pharmacokinetic Analysis Set (PKS) | 260 | 258 | 0 | 0 | 0
TP1 Safety Analysis Set | 263 | 264 | 0 | 0 | 0
Completed | 253 | 249 | 0 | 0 | 0
Not Completed | 10 | 15 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Not completed — Subject decision | 8 | 9 | 0 | 0 | 0
Period: TP2- Week 52 to Week 78
Arm/Group | GP2411 | EU-Prolia | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Started | 0 | 0 | 253 | 125 | 124
TP2 Full Analysis Set (TP2 FAS) | 0 | 0 | 253 | 124 | 124
TP2 Safety Analysis Set | 0 | 0 | 253 | 125 | 124
Completed | 0 | 0 | 253 | 123 | 124
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Subject decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2411 | EU-Prolia | Total
Number analyzed (Participants) | 263 | 264 | 527
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (6.08) | 64.7 (5.78) | 64.7 (5.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 264 | 527
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 23 | 24 | 47
  Multiple | 1 | 0 | 1
  White | 239 | 240 | 479

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 52 - Per-Protocol Set
Description: Bone density measurements were performed by dual energy X-ray absorptiometry (DXA). Lumbar spine scan included L1 through L4 vertebrae. All DXA scans were submitted to a central imaging vendor for analysis. A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in LS-BMD for all post-baseline time points up to Week 52. Values at Week 52 were estimated from the model and are presented in the table.
Time Frame: Baseline (screening), up to Week 52
Population: Per-Protocol Set (PPS) defined as participants who were randomized into TP1 and met the following criteria: the LS-BMD assessments at baseline and Week 52 are available, they received treatment according to protocol on Day 1 and Week 26 and they did not experience relevant protocol deviations which would affect LS-BMD up to Week 52.
Measure: Least Squares Mean (Standard Error); unit: Percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 233 | 230
Percentage change (%) | 4.955 (0.2634) | 5.099 (0.2618)
Statistical Analysis 1: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set PPS): 95% CI for difference in means contained in [-1.45%, 1.45%]; Mixed-model repeated measures (MMRM); MMRM included treatment, prior bisphosphonate use, DXA machine type, visit, visit-treatment interaction, and baseline LS-BMD as a continuous covariate; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.798 to 0.509], Standard Error of Mean 0.3325 — Difference GP2411 (Test) - EU-Prolia (Reference)

2. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 52 - TP1 Full Analysis Set
Description: Bone density measurements were performed by DXA. Lumbar spine scan included L1 through L4 vertebrae. All DXA scans were submitted to a central imaging vendor for analysis. A MMRM was fitted to the changes from baseline in LS-BMD for all post-baseline time points up to Week 52. Missing values were assumed to be missing at random (MAR) using the MMRM model. Values at Week 52 were estimated from the model and are presented in the table.
Time Frame: Baseline (screening), up to Week 52
Population: TP1 Full Analysis Set (TP1 FAS) defined as participants who were randomized into TP1, who received at least one dose of study drug and for whom at least one post-baseline LS-BMD value (either at Week 26 or Week 52 or at both visits) is available.
Measure: Least Squares Mean (Standard Error); unit: Percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 255 | 257
Percentage change (%) | 4.963 (0.2630) | 5.140 (0.2627)
Statistical Analysis 1: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set TP1 FAS): 95% CI for difference in means contained in [-1.45%, 1.45%] (criteria 1) or in [-2.00%, 2.00%] (criteria 2); Mixed-model repeated measures (MMRM); [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.177, 95% CI 2-sided [-0.830 to 0.475], Standard Error of Mean 0.3321 — Difference GP2411 (Test) - EU-Prolia (Reference)

3. Primary Outcome: Area Under the Effect-time Curve (AUEC) of Percentage Change From Baseline in Serum CTX Concentrations After First Dose - Pharmacodynamic Analysis Set
Description: Carboxy-terminal crosslinked telopeptides of type I collagen (CTX) is a bone resorption biomarker. Serum CTX concentration-time data were analyzed by non-compartmental methods. The AUEC of baseline corrected serum CTX concentrations (% change from baseline) was calculated using the linear trapezoidal method. Values below the lower limit of quantification (LLOQ) were imputed with the actual value for the LLOQ.
Time Frame: Baseline (pre-dose Day 1), up to Week 26
Population: Pharmacodynamic Analysis Set (PDS) defined as participants who were randomized into TP1 and met the following criteria: CTX values are available in order to be able to calculate AUEC, they received treatment according to protocol on Day 1 and they did not experience relevant protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage change (%)*day
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 228 | 213
percentage change (%)*day | 15700 (15.8) | 15900 (14.0)
Statistical Analysis 1: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set PDS): 95% CI for ratio of geometric means contained in [0.80, 1.25%]; ANCOVA; ANCOVA was performed on log-transformed AUEC including treatment and log baseline CTX value as a continuous covariate; Geometric mean ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — Geometric mean ratio of GP2411 (Test) to EU-Prolia (Reference)
Statistical Analysis 2: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set PDS): 90% CI for ratio of geometric means contained in [0.80, 1.25%]; ANCOVA; ANCOVA was performed on log-transformed AUEC including treatment and log baseline CTX value as a continuous covariate; Geometric mean ratio = 1.00, 90% CI 2-sided [0.98 to 1.01] — Geometric mean ratio of GP2411 (Test) to EU-Prolia (Reference)

4. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Denosumab After First Dose
Description: Serum denosumab concentration-time data were analyzed by non-compartmental methods. Missing denosumab serum concentrations or concentrations below the LLOQ were not imputed and handled as missing values, except for the pre-dose sample which were treated as zero.
Time Frame: Baseline (pre-dose Day 1), up to Week 26
Population: Participants in the Pharmacokinetic Analysis Set (PKS) who had valid assessments of Cmax. The PKS is defined as participants who were randomized into TP1 and met the following criteria: at least one PK primary endpoint (Cmax or AUCinf) is evaluable, they received treatment according to protocol on Day 1 and they did not experience relevant protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 260 | 258
ng/mL | 6970 (45.8) | 7050 (44.2)
Statistical Analysis 1: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set PKS): 90% CI for ratio of geometric means contained in [0.80, 1.25%]; ANCOVA; ANCOVA was performed on log-transformed Cmax including treatment and weight as a continuous covariate; Geometric mean ratio = 0.97, 90% CI 2-sided [0.92 to 1.03] — Geometric mean ratio of GP2411 (Test) to EU-Prolia (Reference)

5. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf) of Denosumab After First Dose
Description: Serum denosumab concentration-time data were analyzed by non-compartmental methods. Missing denosumab serum concentrations or concentrations below the LLOQ were not imputed and handled as missing values, except for the pre-dose sample which were treated as zero. The linear-up log-down trapezoidal method was used for the AUCinf calculation.
Time Frame: Baseline (pre-dose Day 1), up to Week 26
Population: Participants in the Pharmacokinetic Analysis Set (PKS) who had valid assessments of AUCinf. The PKS is defined as participants who were randomized into TP1 and met the following criteria: at least one PK primary endpoint (Cmax or AUCinf) is evaluable, they received treatment according to protocol on Day 1 and they did not experience relevant protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 247 | 246
day*ng/mL | 370000 (47.8) | 365000 (43.3)
Statistical Analysis 1: Comparison: GP2411 vs EU-Prolia; Test type: Equivalence — Equivalence criteria (analysis set PKS): 90% CI for ratio of geometric means contained in [0.80, 1.25%]; ANCOVA; ANCOVA was performed on log-transformed AUCinf including treatment and weight as a continuous covariate; Geometric mean ratio = 0.99, 90% CI 2-sided [0.93 to 1.05] — Geometric mean ratio of GP2411 (Test) to EU-Prolia (Reference)

6. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 26 - Treatment Period 1 (Per-Protocol Set)
Description: Bone density measurements were performed by DXA. Lumbar spine scan included L1 through L4 vertebrae. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Week 26
Population: Participants in the Per-Protocol Set (PPS) who had valid assessments of the outcome measure at both baseline and Week 26.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 233 | 229
percentage change (%) | 3.6501 (3.76952) | 3.6700 (3.68816)

7. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 26 - Treatment Period 1 (TP1 Full Analysis Set)
Description: as for outcome 6
Time Frame: Baseline (screening), Week 26
Population: Participants in the TP1 Full Analysis Set (TP1 FAS) who had valid assessments of the outcome measure at both baseline and Week 26.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 255 | 256
percentage change (%) | 3.5877 (3.73579) | 3.7144 (3.89730)

8. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (LS-BMD) at Week 78 - Treatment Period 2 (TP2 Full Analysis Set)
Description: Bone density measurement were performed by DXA. Lumbar spine scan included L1 through L4 vertebrae. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Week 78
Population: Participants in the TP2 Full Analysis Set (TP2 FAS) who had valid assessments of the outcome measure at both baseline and Week 78. TP2 FAS is defined as participants who were re-randomized into TP2 and for whom at least one TP2 efficacy, pharmacokinetics or pharmacodynamics value is available.
Measure: Mean (Standard Deviation); unit: Percentage change (%)
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 249 | 123 | 122
Percentage change (%) | 6.8222 (3.95225) | 7.0694 (4.72955) | 6.4212 (4.47102)

9. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (FN-BMD) at Week 26 and Week 52 - Treatment Period 1 (Per-Protocol Set)
Description: Bone density measurements were performed by DXA. For proximal femur, the left side was to be used for all DXA scans at all study visits. If the right side had to be used (e.g., due to implants) or was inadvertently used at baseline, then it was to be used consistently throughout the study. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Week 26 and Week 52
Population: The overall number of participants analyzed represents the Per-Protocol Set (PPS). The number analyzed per row represents participants with data at baseline and at the corresponding time point.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 233 | 230
percentage change (%)
  Week 26: number analyzed (Participants) | 232 | 229
  Week 26 | 2.0818 (3.38039) | 1.8087 (3.18505)
  Week 52: number analyzed (Participants) | 233 | 229
  Week 52 | 2.4200 (3.70552) | 2.6157 (3.26119)

10. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (FN-BMD) at Week 26 and Week 52 - Treatment Period 1 (TP1 Full Analysis Set)
Description: as for outcome 9
Time Frame: Baseline (screening), Week 26 and Week 52
Population: The overall number of participants analyzed represents the TP1 Full Analysis Set (TP1 FAS). The number analyzed per row represents participants with data at baseline and at the corresponding time point.
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 255 | 257
percentage change (%)
  Week 26: number analyzed (Participants) | 254 | 256
  Week 26 | 2.0343 (3.43682) | 1.8210 (3.11073)
  Week 52: number analyzed (Participants) | 253 | 248
  Week 52 | 2.3686 (3.69145) | 2.5717 (3.29726)

11. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (FN-BMD) at Week 78 - Treatment Period 2 (TP2 Full Analysis Set)
Description: as for outcome 9
Time Frame: Baseline (screening), Week 78
Population: Participants in the TP2 Full Analysis Set (TP2 FAS) who had valid assessments of the outcome measure at both baseline and Week 78.
Measure: Mean (Standard Deviation); unit: Percentage change (%)
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 247 | 122 | 122
Percentage change (%) | 3.2220 (4.03733) | 2.9406 (3.92115) | 2.6857 (3.64193)

12. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (TH-BMD) at Week 26 and Week 52 - Treatment Period 1 (Per-Protocol Set)
Description: Bone density measurements were performed by DXA. For total hip, the left side was to be used for all DXA scans at all study visits. If the right side had to be used (e.g., due to implants) or was inadvertently used at baseline, then it was to be used consistently throughout the study. All DXA scans were submitted to a central imaging vendor for analysis.
Time Frame: Baseline (screening), Week 26 and Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 233 | 230
percentage change (%)
  Week 26: number analyzed (Participants) | 232 | 229
  Week 26 | 2.6475 (2.43928) | 2.1178 (2.44627)
  Week 52: number analyzed (Participants) | 233 | 229
  Week 52 | 3.4289 (2.71152) | 3.3211 (2.59266)

13. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (TH-BMD) at Week 26 and Week 52 - Treatment Period 1 (TP1 Full Analysis Set)
Description: as for outcome 12
Time Frame: Baseline (screening), Week 26 and Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change (%)
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 255 | 257
percentage change (%)
  Week 26: number analyzed (Participants) | 254 | 256
  Week 26 | 2.5280 (2.46669) | 2.0595 (2.51811)
  Week 52: number analyzed (Participants) | 253 | 248
  Week 52 | 3.2882 (2.70260) | 3.2234 (2.64633)

14. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (TH-BMD) at Week 78 - Treatment Period 2 (TP2 Full Analysis Set)
Description: Bone density measurements were performed by DXA. For total hip, the left side was to be used for all DXA scans at all study visits. If the right side had to be used (e.g., due to implants) or was inadvertently used at baseline, then it was to be used consistently throughout the study.
Time Frame: Baseline (screening), Week 78
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage change (%)
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 247 | 122 | 122
Percentage change (%) | 3.8270 (3.28071) | 4.0898 (2.96530) | 3.9987 (3.33311)

15. Secondary Outcome: CTX Serum Concentrations as Per Visit Schedule up to Week 52 - Treatment Period 1
Description: CTX is a bone resorption biomarker. Serum samples were analyzed for CTX concentrations. CTX serum concentrations were determined by a validated ligand-binding immunoassay. Values below the LLOQ were imputed with the actual value for the LLOQ.
Time Frame: Baseline (pre-dose Day 1), Day 2, Day 4, Week 8, Week 18, Week 22, Week 26, Week 39 and Week 52
Population: The overall number of participants analyzed represents the Pharmacodynamic Analysis Set (PDS). The number analyzed per row represents participants with data at the corresponding time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 228 | 213
ng/mL
  Baseline | 0.437 (0.249) | 0.450 (0.264)
  Day 2: number analyzed (Participants) | 226 | 212
  Day 2 | 0.0904 (0.110) | 0.0859 (0.0923)
  Day 4: number analyzed (Participants) | 226 | 211
  Day 4 | 0.0383 (0.0272) | 0.0407 (0.0537)
  Week 8: number analyzed (Participants) | 222 | 206
  Week 8 | 0.0339 (0.0134) | 0.0332 (0.00334)
  Week 18: number analyzed (Participants) | 219 | 200
  Week 18 | 0.0355 (0.0205) | 0.0362 (0.0225)
  Week 22: number analyzed (Participants) | 226 | 211
  Week 22 | 0.0428 (0.0546) | 0.0422 (0.0406)
  Week 26 | 0.0661 (0.0954) | 0.0651 (0.0708)
  Week 39: number analyzed (Participants) | 227 | 206
  Week 39 | 0.0342 (0.0116) | 0.0345 (0.0110)
  Week 52: number analyzed (Participants) | 224 | 207
  Week 52 | 0.0845 (0.116) | 0.0807 (0.0883)

16. Secondary Outcome: CTX Serum Concentrations as Per Visit Schedule From Week 52 up to Week 78 - Treatment Period 2
Description: as for outcome 15
Time Frame: Week 56, Week 65 and Week 78
Population: The overall number of participants analyzed represents the TP2 Full Analysis Set (TP2 FAS). The number analyzed per row represents participants with data at the corresponding time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 124 | 124
ng/mL
  Week 56: number analyzed (Participants) | 247 | 116 | 117
  Week 56 | 0.0335 (0.00685) | 0.0358 (0.0259) | 0.0330 (0.00)
  Week 65: number analyzed (Participants) | 246 | 117 | 118
  Week 65 | 0.0335 (0.00714) | 0.0352 (0.0159) | 0.0359 (0.0281)
  Week 78: number analyzed (Participants) | 248 | 117 | 117
  Week 78 | 0.125 (0.190) | 0.144 (0.155) | 0.101 (0.149)

17. Secondary Outcome: PINP Serum Concentrations as Per Visit Schedule up to Week 52 - Treatment Period 1
Description: Procollagen I N-terminal propeptide (PINP) is a bone formation biomarker. Serum samples were analyzed for PINP concentrations. PINP serum concentrations were determined by a validated ligand-binding immunoassay. Values below the LLOQ were imputed with the actual value for the LLOQ.
Time Frame: Baseline (pre-dose Day 1), Day 2, Day 4, Week 8, Week 18, Week 22, Week 26, Week 39 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 228 | 213
ng/mL
  Baseline | 60.3 (27.1) | 62.2 (30.0)
  Day 2 | 58.5 (25.9) | 60.2 (29.3)
  Day 4: number analyzed (Participants) | 227 | 213
  Day 4 | 56.8 (23.2) | 58.8 (26.8)
  Week 8: number analyzed (Participants) | 223 | 207
  Week 8 | 21.2 (9.53) | 21.0 (7.58)
  Week 18: number analyzed (Participants) | 221 | 200
  Week 18 | 12.1 (4.52) | 12.6 (5.10)
  Week 22: number analyzed (Participants) | 227 | 212
  Week 22 | 13.5 (5.92) | 13.3 (4.59)
  Week 26 | 15.4 (7.44) | 15.9 (6.71)
  Week 39: number analyzed (Participants) | 227 | 208
  Week 39 | 10.5 (3.14) | 10.7 (3.43)
  Week 52: number analyzed (Participants) | 225 | 207
  Week 52 | 15.0 (5.95) | 15.7 (7.11)

18. Secondary Outcome: PINP Serum Concentrations as Per Visit Schedule From Week 52 up to Week 78 - Treatment Period 2
Description: PINP is a bone formation biomarker. Serum samples were analyzed for PINP concentrations. PINP serum concentrations were determined by a validated ligand-binding immunoassay. Values below the LLOQ were imputed with the actual value for the LLOQ.
Time Frame: Week 56, Week 65 and Week 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 124 | 124
ng/mL
  Week 56: number analyzed (Participants) | 252 | 122 | 124
  Week 56 | 13.7 (8.06) | 13.9 (5.39) | 14.4 (11.0)
  Week 65: number analyzed (Participants) | 250 | 123 | 123
  Week 65 | 10.5 (3.40) | 10.9 (3.43) | 11.1 (3.85)
  Week 78: number analyzed (Participants) | 252 | 123 | 124
  Week 78 | 17.5 (14.1) | 20.3 (20.4) | 17.1 (8.37)

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs up to Week 52 - Treatment Period 1
Description: Number of participants with TEAEs and serious TEAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs during Treatment Period 1.
  The number of participants in each category is reported in the table.
Time Frame: From first dose of study treatment on Day 1 up to pre-dose at Week 52
Population: TP1 Safety Analysis Set defined as participants who received at least one dose of study drug in Treatment Period 1.
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 263 | 264
Participants
  TEAE | 157 | 181
  Treatment-related TEAE | 36 | 49
  Serious TEAE | 12 | 8
  Treatment-related serious TEAE | 0 | 0

20. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs From Week 52 up to Week 78 - Treatment Period 2
Description: Number of participants with TEAEs and serious TEAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs during Treatment Period 2.
  The number of participants in each category is reported in the table.
Time Frame: From dosing of study treatment at Week 52 up to Week 78
Population: TP2 Safety Analysis Set defined as participants who received at least one dose of study drug in Treatment Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 125 | 124
Participants
  TEAE | 68 | 47 | 48
  Treatment-related TEAE | 7 | 7 | 5
  Serious TEAE | 4 | 2 | 0
  Treatment-related serious TEAE | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Vertebral Fractures up to Week 52 - Treatment Period 1
Description: Vertebral fractures were assessed by independent radiologists at the central imaging vendor. The radiologists assessed lateral thoracic (vertebrae T4 to T12) and lumbar (vertebrae L1 to L4) spine radiographs for vertebral fractures. New and worsening vertebral fractures are defined as occurrence of new fracture (i.e. change in Genant score from 0 at baseline to 1 or higher at a later time point) or worsening fracture (i.e. increase in Genant score from baseline at a later time point) in any assessed vertebra. The Genant classification of vertebral fractures is based on the vertebral shape, with respect to vertebral height loss involving the anterior, posterior, and/or middle vertebral body and ranges between 0 (normal) and 3 (severe fracture, >40% loss of height).
  The number of participants in each category is reported in the table.
Time Frame: Baseline (screening) and Week 52
Population: All participants in the TP1 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 263 | 264
Participants
  At least one vertebral fracture at baseline | 123 | 116
  New vertebral fractures at Week 52 | 15 | 24
  Worsening vertebral fractures at Week 52 | 3 | 3

22. Secondary Outcome: Number of Participants With Vertebral Fractures From Week 52 up to Week 78 - Treatment Period 2
Description: Vertebral fractures were assessed by independent radiologists at the central imaging vendor. The radiologists assessed lateral thoracic (vertebrae T4 to T12) and lumbar (vertebrae L1 to L4) spine radiographs for vertebral fractures. New and worsening vertebral fractures are defined as occurrence of new fracture (i.e. change in Genant score from 0 at Week 52 to 1 or higher at a later time point) or worsening fracture (i.e. increase in Genant score from Week 52 at a later time point) in any assessed vertebra. The Genant classification of vertebral fractures is based on the vertebral shape, with respect to vertebral height loss involving the anterior, posterior, and/or middle vertebral body and ranges between 0 (normal) and 3 (severe fracture, >40% loss of height).
  The number of participants in each category is reported in the table.
Time Frame: Week 52 and Week 78
Population: All participants in the TP2 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 125 | 124
Participants
  At least one vertebral fracture at Week 52 | 126 | 57 | 65
  New vertebral fractures at Week 78 | 12 | 3 | 8
  Worsening vertebral fractures at Week 78 | 1 | 0 | 0

23. Secondary Outcome: Number of Participants With Nonvertebral Fractures up to Week 52 - Treatment Period 1
Description: Information about any nonvertebral fractures while on study were recorded as adverse events. The diagnosis of nonvertebral fractures did not require central X-ray reading and was based on local radiology reports.
  The number of participants in each category is reported in the table.
Time Frame: From first dose of study treatment on Day 1 up to pre-dose at Week 52
Population: All participants in the TP1 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 263 | 264
Participants
  Hip fracture | 2 | 0
  Femoral neck fracture | 1 | 0
  Femur fracture | 0 | 1
  Ankle fracture | 1 | 1
  Wrist fracture | 1 | 0
  Radius fracture | 0 | 1

24. Secondary Outcome: Number of Participants With Nonvertebral Fractures From Week 52 up to Week 78 - Treatment Period 2
Description: as for outcome 23
Time Frame: From dosing of study treatment at Week 52 up to Week 78
Population: All participants in the TP2 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 125 | 124
Participants
  Hip fracture | 1 | 0 | 0
  Fibula fracture | 1 | 0 | 0
  Hand fracture | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) up to Week 52 - Treatment Period 1
Description: The injection site reaction (ISR) assessment was done by the investigator/designee. It consisted of grading the severity of each injection reaction based on criteria the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The ISR grading was defined as follows:
  * Grade 1: Tenderness with or without associated symptoms (e.g., warmth, erythema, itching)
  * Grade 2: Pain; lipodystrophy; edema; phlebitis
  * Grade 3: Ulceration or necrosis; severe tissue damage; operative intervention indicated
  * Grade 4: Life-threatening consequences; urgent intervention indicated The number of participants in each category is reported in the table.
Time Frame: From first dose of study treatment on Day 1 up to pre-dose at Week 52
Population: All participants in the TP1 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 263 | 264
Participants
  ISR Grade 1 | 6 | 9
  ISR Grade 2 | 1 | 1
  ISR Grade 3 | 0 | 0
  ISR Grade 4 | 0 | 0

26. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) From Week 52 up to Week 78 - Treatment Period 2
Description: as for outcome 25
Time Frame: From dosing of study treatment at Week 52 up to Week 78
Population: All participants in the TP2 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 125 | 124
Participants
  ISR Grade 1 | 1 | 0 | 0
  ISR Grade 2 | 0 | 0 | 0
  ISR Grade 3 | 0 | 0 | 0
  ISR Grade 4 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) up to Week 52 - Treatment Period 1
Description: Immunogenicity was evaluated in serum. Samples were screened for potential anti-drug antibodies (ADA) and positive screen results were confirmed using a confirmatory assay. For confirmed ADA positive samples, titers were determined. Confirmed ADAs were also analyzed for their neutralization potential. Patient ADA status was defined as follows:
  * ADA Positive: ADA-positive sample at any time point during TP1
  * ADA Positive, Persistent: 'Persistent' indicates a subject experiencing a positive ADA result at the final visit and with at least 2 consecutive positive ADA results
  * ADA Positive, Transient: 'Transient' indicates a subject experiencing positive ADA result but not qualifying as 'Persistent'
  * ADA titer positive: ADA-positive sample with a titer result ≥ 20 ng/mL
  * NAb Positive: ADA-positive sample with presence of neutralizing antibodies (NAb) The number of participants in each category is reported in the table.
Time Frame: From Week 2 up to Week 52
Population: All participants in the TP1 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 263 | 264
Participants
  ADA Positive | 93 | 108
  ADA Positive, Persistent | 7 | 4
  ADA Positive, Transient | 86 | 104
  ADA titer positive | 2 | 2
  NAb positive | 3 | 1

28. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) From Week 52 up to Week 78 - Treatment Period 2
Description: as for outcome 27
Time Frame: From Week 56 up to Week 78
Population: All participants in the TP2 Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 125 | 124
Participants
  ADA Positive | 42 | 26 | 26
  ADA Positive, Persistent | 3 | 3 | 0
  ADA Positive, Transient | 39 | 23 | 26
  ADA titer positive | 0 | 1 | 0
  NAb positive | 1 | 0 | 1

29. Secondary Outcome: Denosumab Serum Concentrations as Per Visit Schedule up to Week 52 - Treatment Period 1
Description: Serum samples were analyzed for concentrations of free denosumab by using a validated ligand binding assay. Briefly, the concentration of free denosumab was determined by binding to coated ligand molecules.
  Denosumab concentrations below the LLOQ were set to zero in order to calculate arithmetic means.
Time Frame: Baseline (pre-dose Day 1), Day 4, Week 1, Week 2, Week 8, Week 14, Week 18, Week 22, Week 26, Week 39 and Week 52
Population: The overall number of participants analyzed represents the Pharmacokinetic Analysis Set (PKS). The number analyzed per row represents participants with data at the corresponding time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411 | EU-Prolia
Number analyzed (Participants) | 260 | 258
ng/mL
  Day 1: number analyzed (Participants) | 256 | 257
  Day 1 | 0.00 (0.00) | 0.928 (14.9)
  Day 4: number analyzed (Participants) | 258 | 258
  Day 4 | 4930 (2530) | 5250 (2660)
  Week 1: number analyzed (Participants) | 259 | 254
  Week 1 | 6820 (3220) | 6890 (3320)
  Week 2: number analyzed (Participants) | 259 | 255
  Week 2 | 6940 (3040) | 6760 (2890)
  Week 8: number analyzed (Participants) | 253 | 251
  Week 8 | 3160 (1500) | 3070 (1510)
  Week 14: number analyzed (Participants) | 250 | 249
  Week 14 | 1130 (740) | 1090 (797)
  Week 18: number analyzed (Participants) | 248 | 241
  Week 18 | 536 (516) | 495 (487)
  Week 22: number analyzed (Participants) | 256 | 254
  Week 22 | 208 (277) | 198 (392)
  Week 26: number analyzed (Participants) | 252 | 253
  Week 26 | 95.9 (415) | 47.9 (114)
  Week 39: number analyzed (Participants) | 250 | 245
  Week 39 | 1490 (902) | 1390 (787)
  Week 52: number analyzed (Participants) | 250 | 244
  Week 52 | 91.9 (186) | 58.3 (126)

30. Secondary Outcome: Denosumab Serum Concentrations as Per Visit Schedule From Week 52 up to Week 78 - Treatment Period 2
Description: as for outcome 29
Time Frame: Week 56, Week 65 and Week 78
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
Number analyzed (Participants) | 253 | 124 | 124
ng/mL
  Week 56: number analyzed (Participants) | 252 | 122 | 124
  Week 56 | 6010 (2200) | 5550 (1900) | 6220 (2130)
  Week 65: number analyzed (Participants) | 250 | 123 | 122
  Week 65 | 1540 (880) | 1330 (753) | 1640 (962)
  Week 78: number analyzed (Participants) | 251 | 123 | 124
  Week 78 | 122 (406) | 53.2 (133) | 147 (652)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment on Day 1 up to Week 78.
Description: Any sign or symptom that occurs from first dose of study treatment up to 26 weeks after last dose in each treatment period.
Arm/Group | GP2411 | EU-Prolia | GP2411/GP2411 | EU-Prolia/EU-Prolia | EU-Prolia/GP2411
All-Cause Mortality (participants affected / at risk) | 1/263 | 0/264 | 0/253 | 0/125 | 0/124
Serious Adverse Events (participants affected / at risk) | 12/263 | 8/264 | 4/253 | 2/125 | 0/124
Other Adverse Events (participants affected / at risk) | 89/263 | 119/264 | 33/253 | 29/125 | 24/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GP2411 (N=263) | EU-Prolia (N=264) | GP2411/GP2411 (N=253) | EU-Prolia/EU-Prolia (N=125) | EU-Prolia/GP2411 (N=124)
Epiretinal membrane (Eye disorders) | 0 | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GP2411 (N=263) | EU-Prolia (N=264) | GP2411/GP2411 (N=253) | EU-Prolia/EU-Prolia (N=125) | EU-Prolia/GP2411 (N=124)
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 1 | 4 | 0
Injection site reaction (General disorders) | 7 | 10 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 9 | 13 | 6 | 7 | 2
Cystitis (Infections and infestations) | 1 | 9 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 23 | 16 | 5 | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 5 | 10 | 2 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 6 | 1 | 1 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 5 | 2 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 28 | 26 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 12 | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 8 | 7 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 2 | 2 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 9 | 0 | 2 | 1
Headache (Nervous system disorders) | 6 | 13 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03974100/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03974100/SAP_001.pdf